CLINICAL TRIAL: NCT02839252
Title: Iggy and the Inhalers: A Pilot Study to Assess the Impact of an Asthma Education Program in School Age Children
Brief Title: Iggy and the Inhalers: A Study to Assess the Impact of an Asthma Education Program in School Age Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6404
Record Dates: First submitted 2016-07-15; First posted 2016-07-20 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2018-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (2):
- Intervention Group (Experimental): After the baseline tools have been completed, the child will be given the Iggy Comic Book and trading cards. Parents and their children will then watch a 12-minute Iggy Video. At the completion of the video and prior to going home, the child and parent will complete the same 2 measures on asthma knowledge and self-efficacy. At 1-month after this clinic visit, the parent will be sent an email with a link to a Qualtrics survey that will contain a few supplemental questions to assess use of the intervention and the same 2 measures that the parent and the child completed at the initial visit.
  Interventions: Behavioral: Iggy and the Inhalers Asthma Education for Kids
- Control Group (No Intervention): After the baseline tools have been completed, the parent and child will go home. At 1-month after the initial study clinic visit, the parent will be sent an email with a link to a Qualtrics survey that will contain a few supplemental questions to assess use of the intervention and the same 2 measures that the parent and the child completed at the initial visit.

INTERVENTIONS:
Behavioral: Iggy and the Inhalers Asthma Education for Kids — It is a comic book, trading cards, and stickers that teach kids about asthma. There is also a 12-minute cartoon video which teaches kids about asthma.
  Arms: Intervention Group

SUMMARY:
The specific aims of this pilot study are to:

1. Evaluate the effectiveness of the asthma education intervention on asthma knowledge
2. Determine whether the asthma education intervention improves child and parent asthma treatment self-efficacy

Our hypothesis is that the asthma education intervention will significantly improve asthma knowledge and asthma self-efficacy at 1 month post-intervention as compared to controls.

DETAILED DESCRIPTION:
Potential subjects will be recruited from patients seen at Yacktman General Pediatrics Clinic. Investigators will initially use the clinic's electronic medical record (EMR) to identify potentially eligible subjects who have a regularly scheduled visit during the next 4 months. Once the patient is deemed eligible, they will be marked as "ASTHMA STUDY ELIGIBLE" in a red banner in the EMR. The parent will then be mailed a recruitment letter with parent permission/consent and child assent forms attached for their review. Once a potentially eligible patient shows up for a sick visit or a well visit, they will receive a handout reminding them of the study and asking them to consider participation. After their clinic visit, a designated pediatric resident will obtain parent permission/consent and child assent. Designated residents are those 2nd and 3rd year pediatric residents who have completed appropriate CITI training and financial conflict of interest disclosure, and have been trained by the PI on the study.

Study Endpoints:

The primary endpoint in this study is asthma knowledge at 2 time points: Immediately after the intervention (at the end of the initial clinic visit) and at 1-month post-intervention.

The secondary endpoint is asthma self-efficacy at the same 2 time points.

Procedures Involved:

This will be a prospective, randomized controlled clinical trial of an asthma educational intervention. It will compare two groups of children and their parents. One cohort will receive the asthma education intervention "Iggy and the Inhalers," and the other cohort will receive usual care in the outpatient, general pediatric clinic setting.

After recruitment procedures have been completed and the child and parent come into clinic for their scheduled visit, a member of the study team (designated resident or PI) will meet them and bring them to a specially designated room in the clinic. This process will occur after the patient's regularly scheduled visit. The study team member will then review the study, answer any questions, and obtain parent permission/consent and child assent. The study team member will indicate enrollment in the EMR by changing the banner to either "ASTHMA STUDY DECLINED" or "ASTHMA STUDY ENROLLED." For those who agree to participate, the parent and child will each be given 2 tools to complete:

* Parent:

  * Asthma Knowledge: Parent Questionnaire
  * Parent Asthma Self-efficacy survey
* Child:

  * Asthma Knowledge: Child Questionnaire
  * Child Self-efficacy Survey

In addition the parent will complete a demographic survey. While they are completing these tools, the study team member will determine the child's group assignment by consulting a random assignment log maintained at the clinic. Randomization will occur in blocks of 10 to allow equal group sizes for interim analyses. After the tools have been completed and collected, the child and parent will be informed of their group assignment, and study procedures will continue as follows.

Intervention Group:

After the baseline tools have been completed, the child will be given the Iggy Comic Book and trading cards. Parents and their children will then watch a 12-minute Iggy Video. At the completion of the video and prior to going home, the child and parent will complete the same 2 measures on asthma knowledge and self-efficacy. At 1-month after this clinic visit, the parent will be sent an email with a link to a Qualtrics survey that will contain a few supplemental questions to assess use of the intervention and the same 2 measures that the parent and the child completed at the initial visit. If we do not receive the completed surveys within 1-2 weeks, we will call them to remind them and offer them over the phone completion. If the parent asks to complete the online surveys they will again be given another 1-2 weeks. If the surveys are still not received, then we will make a 2nd call to repeat this process. If no success after this attempt, they will be deemed lost to follow-up. Once the surveys have been completed or the parent/child are deemed lost to follow up, the outpatient EMR banner will be changed to "ASTHMA STUDY COMPLETE." When the parent and child complete the final surveys, a thank you letter will be sent to the child and parent.

Control Group:

After the baseline tools have been completed, the parent and child will go home. At 1-month after the initial study clinic visit, the parent will be sent an email with a link to a Qualtrics survey that will contain a few supplemental questions to assess use of the intervention and the same 2 measures that the parent and the child completed at the initial visit. If the study team does not receive the completed surveys within 1-2 weeks, investigators will call them to remind them and offer them over the phone completion. If the parent asks to complete the online surveys the parents and children will again be given another 1-2 weeks. If the surveys are still not received, then investigators will make a 2nd call to repeat this process. If no success after this attempt, will be deemed lost to follow-up. Once the surveys have been completed or the parent/child are deemed lost to follow up, the outpatient EMR banner will be changed to "ASTHMA STUDY COMPLETE." When the parent and child complete the final surveys, the PI will send the control group a thank you letter with Iggy Comic Book, trading cards, and link to Iggy videos included.

Measures / Data Collection:

* Demographic Survey

  o Includes: age, gender, ethnicity/race, primary language, residential zip code, education level of caregiver, annual household income, # of ED visits/hospitalizations for asthma symptoms over the past 1year. Baseline demographic information will be collected for each parent and child during the initial visit. These baseline measures include background information, which could become possible confounders for the study. This information is based on background information from similar studies published in this area.
* Asthma Knowledge Test Parent/Child

  o Asthma knowledge will be assessed using 10-item multiple-choice questionnaires for both parents and children that was developed by Butz et al. Content was derived from the current National Asthma Educational Prevention Program (NAEPP) Guidelines, asthma symptom identification interventions, and was derived from a prior study on asthma education with the original authors permission. The child form was used in children 6-12 years of age. The final 10-item Asthma Knowledge Questionnaire reading level was written at a 4.7 grade level (Flesch-Kincaid grade level). Content validity of the parent and child knowledge scales, were assessed by an expert panel of pediatric allergists and general pediatricians, was high. Total scores on the asthma knowledge scale range from 0 to 10 points.
* Asthma Management Self-Efficacy Survey Parent/Child

  o Self-efficacy will be assessed using a 13-question (Parent) and a 14-question (Child) survey. The survey utilizes a Likert scale response format and was designed to measure self-efficacy with regard to attack prevention and attack management. Acceptable to very good internal consistency reliabilities (Cronbach's alpha) were obtained for the final measures: Parent Asthma Self-Efficacy (alpha = 0.87) and Child Asthma Self-Efficacy (alpha = 0.87). The Parent Asthma Self-efficacy scale was positively correlated with parent ratings of their child's overall health, parent treatment efficacy, and child asthma self-efficacy. Child Asthma Self-efficacy was positively correlated with parent ratings of their children's health, Parent Asthma Self-Efficacy, Parent Treatment Efficacy, and the age of the child.
* Supplemental Questions to Assess Use of Intervention o These questions will allow us to assess the intervention dose. They will also provide feedback on the education program and allow it to be tailored to different pediatric populations.

Data to be recorded:

* Demographics (age, gender, ethnicity, primary language, residential zip code, education level of child and caregiver, household income, # of ED visits/hospitalizations for asthma symptoms over the past 1year)
* Asthma Knowledge Test Parent/Child: pre-, post-, and 1-month follow up scores
* Self Efficacy Survey Parent/Child: pre-, post-, 1-month follow up scores
* Responses to Supplemental Survey to Assess Use of the Intervention
* Comments on the program from parents and patients

ELIGIBILITY:
Inclusion Criteria:

* Followed in the Yacktman General Pediatrics Clinic at Advocate Children's Hospital - Park Ridge (ACH-PR)
* Age 8 - 12 years
* Documented diagnosis of asthma (any severity level)
* Child and parent are English-speaking
* Child is currently taking an asthma medication on either a daily or an as-needed basis
* Parent permission/consent and child assent is obtained

Exclusion Criteria:

* Child has a diagnosis of another chronic lung or cardiovascular disease
* Child was assessed by parents or clinician to have a significant developmental delay, learning, or behavioral disability (e.g., autism spectrum)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Asthma knowledge | Change in asthma knowledge immediately post-intervention and 1 month after intervention as compared with asthma knowledge prior to the intervention
  This will be measured by a 10 question multiple choice survey

SECONDARY OUTCOMES:
Asthma Self Efficacy | Change in asthma self efficacy scores immediately post-intervention and 1 month after intervention as compared to pre-intervention self-efficacy scores
  This will be measured by a 14 question survey

CONTACTS AND LOCATIONS:
Locations (1):
- Yacktman Pediatrics, Park Ridge, Illinois, United States